CLINICAL TRIAL: NCT00443898
Title: A Randomized, Double-blind, Vehicle-controlled, Multicenter, Parallel Group Study to Assess the Efficacy, Safety, and Tolerability of Topical Terbinafine Hydrogen Chloride (HCl) Formulation for 24 or 48 Weeks of Treatment in Patients With Mild to Moderate Toenail Onychomycosis
Brief Title: Efficacy, Safety, and Tolerability of Topical Terbinafine in Patients With Mild to Moderate Toenail Fungus of the Big Toenail
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSFO327N2301
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Onychomycosis
Keywords: Toenail fungus; Onychomycosis; Nail fungus; Toenail fungal infection; Tinea unguium; Dermatophytes; Foot dermatoses
MeSH Terms: conditions — Onychomycosis; Foot Dermatoses | interventions — Terbinafine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Active terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) applied once daily for 48 weeks
  Interventions: Drug: terbinafine
- 2 (Placebo Comparator): vehicle (placebo) applied once daily for 48 weeks
  Interventions: Drug: Placebo
- 3 (Experimental): Active terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) applied once daily for 24 weeks
  Interventions: Drug: terbinafine
- 4 (Placebo Comparator): vehicle (placebo) applied once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: terbinafine — Active terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) once daily for 48 weeks
  Other Names: Lamisil
  Arms: 1
Drug: Placebo — vehicle (placebo) applied once daily for 48 weeks
  Arms: 2
Drug: terbinafine — Active terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) once daily for 24 weeks
  Other Names: Lamisil
  Arms: 3
Drug: Placebo — vehicle (placebo) applied once daily for 24 weeks
  Arms: 4

SUMMARY:
This study is designed to assess the efficacy, safety and tolerability of a topical formulation of terbinafine solution applied daily in patients with toenail fungus. This trial will study patients with mild to moderate toenail fungus disease of the big toenail and their responses to two treatment durations, 24 or 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 12 - 75 years of age
* Fungal toenail infection of one or both of the large (great) toenails
* The nail infection must be due to a dermatophyte, (mixed infections [dermatophyte and non-dermatophyte] are not allowed)

Exclusion Criteria:

* Target foot must not have severe plantar (moccasin) tinea pedis that would require systemic therapy. Mild to moderate tinea pedis (athlete's foot) infection should be treated with terbinifine prior to baseline or at any time during the trial. Other topical treatments for athlete's foot may be recommended at the discretion of the investigator.
* Subjects must not have abnormalities of the nail that could prevent a normal appearing nail if clearing of infection is achieved
* No administration of systemic antifungal medications within 6 months prior to screening visit
* No application of prescription topical antifungal medications for toenail fungus within 3 months or other commercially available topical medications for toenail fungus applied directly to the toenails within 1 month prior to screening visit
* No professional pedicures or application of any nail polish product or nail cosmetic to the toenails after the screening visit
* Known pregnancy or lactation at time of enrollment

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (20):
  - Dr. Boni Elewski, Birmingham, Alabama
  - Dr. Stacy Smith, San Diego, California
  - Dr. James Swinehart, Denver, Colorado
  - Dr. David G. Armstrong, North Chicago, Illinois
  - Dr. Kevin Terry, Lutherville, Maryland
  - Dr. Anthony Puopolo, Milford, Massachusetts
  - Dr. John Fenyk, Chaska, Minnesota
  - Dr. Joel Schlessinger, Omaha, Nebraska
  - Dr. AnneMarie Uliasz, New York, New York
  - Dr. Willard Niemi, Raleigh, North Carolina
  - Dr. Diane Baker, Lake Oswego, Oregon
  - Dr. John Barnes, Portland, Oregon
  - Dr. Harry Penny, Altoona, Pennsylvania
  - Dr. Lawrence Parish, Philadelphia, Pennsylvania
  - Dr. Cynthia Strout, Mt. Pleasant, South Carolina
  - Dr. Teresa Coats, Austin, Texas
  - Dr. Scott J. Ashton, Dallas, Texas
  - Dr. Amit Pandya, Dallas, Texas
  - Dr. Lawrence Harkless, San Antonio, Texas
  - Dr. Robert Shouey, Harrisonburg, Virginia
- Novartis Investigative Site, Various Cities, Canada
- Novartis Investigative Site, Various Cities, Iceland

RESULTS

PARTICIPANT FLOW:
Groups:
- Terbinafine 24 w: Active terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) applied once daily for 24 weeks
- Vehicle 24 w: vehicle (placebo) applied once daily for 24 weeks
- Terbinafine 48 w: Active terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) applied once daily for 48 weeks
- Vehicle 48 w: vehicle (placebo) applied once daily for 48 weeks
Period: Overall Study
Arm/Group | Terbinafine 24 w | Vehicle 24 w | Terbinafine 48 w | Vehicle 48 w
Started | 126 | 128 | 136 | 128
Completed | 102 | 103 | 107 | 110
Not Completed | 24 | 25 | 29 | 18
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 2 | 3 | 3 | 1
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 10 | 10 | 6
Not completed — Lost to Follow-up | 10 | 10 | 14 | 10
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terbinafine 24 w | Vehicle 24 w | Terbinafine 48 w | Vehicle 48 w | Total
Number analyzed (Participants) | 126 | 128 | 136 | 128 | 518
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 107 | 101 | 116 | 100 | 424
  >=65 years | 19 | 27 | 20 | 28 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 26 | 27 | 107
  Male | 101 | 99 | 110 | 101 | 411

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Assessed by Complete Cure Rate at the End of Study (Week 52) After Treating for 24 or 48 Weeks.
Description: Complete cure is defined as negative KOH microscopy and negative culture for dermatophytes.
  and no residual involvement of the target toenail. The complete cure was a composite binary variable defined as "Yes" if:
  * Mycological cure (negative KOH and negative culture for dermatophytes) and
  * No residual involvement of the target toenail "No" if otherwise
Time Frame: 52 weeks
Population: All participants were included in the intention to treat (ITT) population, defined as all participants who were randomized and received study drug. The Last Observation was Carried Forward (LOCF).
Measure: Number; unit: Percentage of Participants
Arm/Group | Terbinafine 24 w | Vehicle 24 w | Terbinafine 48 w | Vehicle 48 w
Number analyzed (Participants) | 126 | 128 | 136 | 128
Percentage of Participants | 0.79 [-2.16 to 2.19] | 0.78 [-2.16 to -2.16] | 1.47 [-0.55 to 3.49] | 0.00 [-0.55 to 3.49]

2. Secondary Outcome: Efficacy Assessed by Mycological Cure (Negative Culture and Negative KOH Microscopy) at the End of Study After Treating Patients for 24 or 48 Weeks.
Description: Mycological cure is defined as negative KOH microscopy and negative culture for dermatophytes.
  Mycological cure was a composite binary variable defined as "Yes"if :
  * Negative microscopy and
  * Negative culture for dermatophytes "No" if otherwise.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Terbinafine 24 w | Vehicle 24 w | Terbinafine 48 w | Vehicle 48 w
Number analyzed (Participants) | 126 | 128 | 136 | 128
Percentage of Participants | 10.32 [-2.70 to 10.83] | 6.25 [-2.70 to 10.83] | 15.44 [5.54 to 19.10] | 3.13 [5.54 to 19.10]

3. Secondary Outcome: Efficacy Assessed by Clinical Efficacy at the End of Study After Treating Patients for 24 or 48 Weeks.
Description: Clinical effectiveness is defined as negative KOH microscopy and negative culture for dermatophytes and <= 10% residual involvement of the target toenail.
  Clinical effectiveness was a composite binary variable defined as "Yes" if
  * Mycological cure (negative KOH and negative culture for dermatophytes) and
  * = 10% residual involvement of the target toenail "No" if otherwise
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Terbinafine 24 w | Vehicle 24 w | Terbinafine 48 w | Vehicle 48 w
Number analyzed (Participants) | 126 | 128 | 136 | 128
Percentage of Participants | 1.59 | 2.34 | 3.68 | 1.56

4. Secondary Outcome: Number of Participants Assessed With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any adverse change in health or side effect that occurs while the participant is receiving the treatment or within a previously specified period of time after the treatment has been completed.
  A Serious Adverse Event (SAE) is any untoward medical occurrence that results in death, is life-threatening requires, inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage.
Time Frame: 52 weeks
Population: Safety Population was defined as all participants who received at least one dose of study drug and had at least one post-baseline safety assessment. All except 4 participants who were randomized to the vehicle 24 w group and one participant randomized to the terbinafine 48 w group, were included in the safety population.
Measure: Number; unit: Participants
Arm/Group | Terbinafine 24 w | Vehicle 24 w | Terbinafine 48 w | Vehicle 48 w
Number analyzed (Participants) | 126 | 124 | 135 | 128
Participants | 126 | 124 | 135 | 128

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Safety Population was defined as all participants who received at least one dose of study drug and had at least one post-baseline safety assessment. All except 4 participants who were randomized to the vehicle 24 w group and one participant randomized to the terbinafine 48 w group, were included in the safety population.
Arm/Group | Terbinafine 24 w | Vehicle 24 w | Terbinafine 48 w | Vehicle 48 w
Serious Adverse Events (participants affected / at risk) | 2/126 | 7/124 | 7/135 | 4/128
Other Adverse Events (participants affected / at risk) | 35/126 | 38/124 | 47/135 | 56/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Terbinafine 24 w (N=126) | Vehicle 24 w (N=124) | Terbinafine 48 w (N=135) | Vehicle 48 w (N=128)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Accidental death (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Terbinafine 24 w (N=126) | Vehicle 24 w (N=124) | Terbinafine 48 w (N=135) | Vehicle 48 w (N=128)
Influenza like illness (General disorders) | 2 | 1 | 0 | 8
Nasopharyngitis (Infections and infestations) | 7 | 9 | 18 | 18
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 9 | 10
Headache (Nervous system disorders) | 23 | 24 | 23 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.